CLINICAL TRIAL: NCT06359678
Title: Assessing the Accuracy of Catheter Localization With NorthStar Software in Real-Time MRI-Guided Cardiac Ablation
Brief Title: The Northstar Trial
Acronym: Northstar
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Luuk Hopman, Principal Investigator, Amsterdam UMC, location VUmc
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL85844.015.23
Record Dates: First submitted 2024-03-18; First posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Flutter, Atrial
MeSH Terms: conditions — Atrial Flutter

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Northstar (Experimental): This is the study group
  Interventions: Device: NorthStar

INTERVENTIONS:
Device: NorthStar — Throughout the real-time MRI-guided ablation procedure, the operator will assess the precision of the NorthStar 3D navigation software. Before commencing the actual ablation, the operator will confirm the alignment of the 3D anatomical shell, generated in NorthStar through specific electrical signals. Post the ablation procedure, a secondary alignment verification will be conducted to detect any potential drift or shift.

SUMMARY:
The introduction of real-time MRI-guided cardiac ablation therapy, a significant advancement in interventional medicine, necessitates precise catheter tracking for accurate navigation within the complex cardiac anatomy. The introduction of the NorthStar software as an active tracking system holds promise for improving the precision and efficiency of catheter manipulation during these procedures. However, a rigorous evaluation of its accuracy and reliability in a clinical setting is crucial to validate its viability.

The objective of this study is to evaluate the accuracy of catheter localization using the NorthStar software during real-time MRI-guided cardiac ablation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a real-time MRI-guided flutter ablation procedure at the Amsterdam UMC.

Exclusion Criteria:

* Lack of legal capacity.
* Insufficient proficiency in the Dutch language.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy of Catheter Localization | during procedure
  The primary objective of this study is to evaluate the accuracy of catheter localization using the NorthStar software during realtime MRI-guided cardiac ablation therapy. At the start of the procedure, the catheters will be manoeuvred to the predefined areas within the right side of the heart based on the specific electrical signals in that area. These locations will be virtually marked within the NorthStar software. The extent to which these markers maintain their spatial coordinates after the ablation procedure, evaluated by obtained electrical signals, will serve as a quantitative measure of the system's accuracy.

SECONDARY OUTCOMES:
Influences of breathing pattern | during procedure
  To investigate the influence of breathing pattern on the accuracy of catheter localization. The breathing pattern during the procedure will be monitored and any changes will be related to the accuracy of catheter localization
Influences of procedure duration | during procedure
  To investigate the influence of procedure duration on the accuracy of catheter localization.
Influences of complications during ablation | during procedure
  To investigate the influence of complications during ablation on the accuracy of catheter localization. Complications during the procedure will be registered and categorized.
Influences of patient characteristics | during procedure
  To investigate the influence of patient characteristics on the accuracy of catheter localization. Standard patient characteristics will be noted such as BMI, cardiac output and heartrate to investigate if these characteristics will influence the catheter localization.

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC, Amsterdam, Netherlands